CLINICAL TRIAL: NCT02419001
Title: A Phase 1b/2a, Randomized, Multi-center, Open-label, Fixed-sequence Study to Evaluate the Effect of Oral SYN-004 on the Pharmacokinetics of Intravenous Ceftriaxone in Healthy Adult Subjects With a Functioning Ileostomy
Brief Title: A Study to Evaluate the Effect of SYN-004 on the PK of IV Ceftriaxone in Adults With a Functioning Ileostomy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theriva Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SB-1-004-003
Record Dates: First submitted 2015-04-01; First posted 2015-04-17 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Period 1 - Treatment Sequence AB (Experimental): Treatment Sequence AB:
  * Period 1: Ceftriaxone 1 g infused IV over 30 minutes
  * [Period 2: Ceftriaxone 1 g infused IV over 30 minutes and SYN-004 75 mg (1 x 75 mg capsule) orally administered 30 minutes before and 5.5 hours after the start of the ceftriaxone infusion]
  Interventions: Drug: Period 1 - Treatment Sequence AB
- Period 1 - Treatment Sequence AC (Experimental): * Period 1: Ceftriaxone 1 g infused IV over 30 minutes
  * [Period 2: Ceftriaxone 1 g infused IV over 30 minutes and SYN-004 150 mg (2 x 75 mg capsules) orally administered 30 minutes before and 5.5 hours after the start of the ceftriaxone infusion]
  Interventions: Drug: Period 1 - Treatment Sequence AC
- Period 2 - Treatment Sequence AB (Experimental): Treatment Sequence AB:
  * [Period 1: Ceftriaxone 1 g infused IV over 30 minutes]
  * Period 2: Ceftriaxone 1 g infused IV over 30 minutes and SYN-004 75 mg (1 x 75 mg capsule) orally administered 30 minutes before and 5.5 hours after the start of the ceftriaxone infusion
  Interventions: Drug: Period 2 - Treatment Sequence AB
- Period 2 - Treatment Sequence AC (Experimental): * [Period 1: Ceftriaxone 1 g infused IV over 30 minutes]
  * Period 2: Ceftriaxone 1 g infused IV over 30 minutes and SYN-004 150 mg (2 x 75 mg capsules) orally administered 30 minutes before and 5.5 hours after the start of the ceftriaxone infusion
  Interventions: Drug: Period 2 - Treatment Sequence AC

INTERVENTIONS:
Drug: Period 1 - Treatment Sequence AB — Period 1: Ceftriaxone 1 g infused IV over 30 minutes only, no SYN-004
  Arms: Period 1 - Treatment Sequence AB
Drug: Period 1 - Treatment Sequence AC — Period 1: Ceftriaxone 1 g infused IV over 30 minutes only, no SYN-004
  Arms: Period 1 - Treatment Sequence AC
Drug: Period 2 - Treatment Sequence AB — Period 2: Ceftriaxone 1 g infused IV over 30 minutes and SYN-004 75 mg
  Other Names: ribaxamase
  Arms: Period 2 - Treatment Sequence AB
Drug: Period 2 - Treatment Sequence AC — Period 2: Ceftriaxone 1 g infused IV over 30 minutes and SYN-004 150 mg
  Other Names: ribaxamase
  Arms: Period 2 - Treatment Sequence AC

SUMMARY:
A Phase 1b/2a, Randomized, Multi-Center, Open-Label, Fixed-Sequence Study to Evaluate the Effect of Oral SYN-004 on the Pharmacokinetics of Intravenous Ceftriaxone in Healthy Adult Subjects with a Functioning Ileostomy.

DETAILED DESCRIPTION:
This is a Phase 1b/2a, randomized, multi-center, open-label study. Twenty otherwise healthy subjects between the ages of 18 and 80 years, inclusive, with functioning ileostomies were planned to be enrolled. In the first treatment period (Period 1) all subjects received an IV infusion of 1 g ceftriaxone. Subjects had a 3 - 7 day washout period between Period 1 and Period 2. In the second treatment period (Period 2) all subjects received an IV infusion of 1 g ceftriaxone and 2 oral doses of either 75 or 150 mg of SYN-004, according to the randomization schedule, which were administered 30 minutes before and 5.5 hours after the start of the ceftriaxone infusion.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a functioning ileostomy which has been in place for > 3 months.
2. Male or female between the ages of 18 and 70 years, inclusive.
3. Other than a functioning ileostomy, the subject is free from clinically significant illnesses or disease.

Exclusion Criteria:

1. Subjects who have active hepatic, small intestine, or biliary tract disease.
2. Subjects who have active ulcerative colitis, Crohn's disease, other inflammatory bowel disease.
3. Subjects with known malignancy requiring treatment < 6 months prior to study screening.
4. Subjects who have, in the opinion of the investigator, significant concurrent medical illness.
5. Subjects who are currently taking concomitant medications which may interfere with study evaluation.
6. Subjects who have received an investigational drug within 30 days or within a time period consistent with a washout period of 5 half-lives, whichever is longer, of the first dose of ceftriaxone.
7. Subjects with a known history of allergy to any cephalosporin, penicillin or any β-lactam antibiotic.
8. Subjects who have known active malabsorption syndromes(s) that, in the judgment of the investigator, could compromise the objectives of the study.
9. Subjects who have used any oral, intramuscular, or IV anti-microbial medication during the last 3 weeks prior to the screening visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kaleko, M.D., Study Chair — Synthetic Biologics
Locations (3):
- Columbus, Ohio, United States
- Canada (2):
  - Edmonton, Alberta
  - Montreal

REFERENCES:
- [Derived] Kokai-Kun JF, Roberts T, Coughlin O, Sicard E, Rufiange M, Fedorak R, Carter C, Adams MH, Longstreth J, Whalen H, Sliman J. The Oral beta-Lactamase SYN-004 (Ribaxamase) Degrades Ceftriaxone Excreted into the Intestine in Phase 2a Clinical Studies. Antimicrob Agents Chemother. 2017 Feb 23;61(3):e02197-16. doi: 10.1128/AAC.02197-16. Print 2017 Mar. PMID 28052855

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose: 1 g ceftriaxone and two low doses (75 mg) of SYN-004
- High Dose: 1 g ceftriaxone and two high doses (150 mg) of SYN-004
Period: Period 1- Ceftriaxone Without SYN-004
Arm/Group | Low Dose | High Dose
Started | 6 | 5
Completed | 5 (The Adverse Event (AE) was with ceftriaxone, not with Investigational Product (IP)) | 5
Not Completed | 1 | 0
Not completed — AE w/ ceftriaxone, not dosed w/ IP | 1 | 0
Period: Period 2- Ceftriaxone With SYN-004
Arm/Group | Low Dose | High Dose
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose: 1 g ceftriaxone and two low doses of SYN-004
- High Dose: 1 g ceftriaxone and two high doses of SYN-004
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.9) | 57.1 (11.6) | 48.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Ceftriaxone PK Maximum Observed Plasma Concentration (Cmax) With (Period 2) and Without (Period 1) SYN-004.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Treatment Sequence AB: Period 1: Ceftriaxone 1 g infused IV over 30 minutes Period 2: Ceftriaxone 1 g infused IV over 30 minutes and SYN-004 75 mg (1 x 75 mg capsule) orally administered 30 minutes before and 5.5 hours after the start of the ceftriaxone infusion
- Treatment Sequence AC: Period 1: Ceftriaxone 1 g infused IV over 30 minutes Period 2: Ceftriaxone 1 g infused IV over 30 minutes and SYN-004 150 mg (2 x 75 mg capsules) orally administered 30 minutes before and 5.5 hours after the start of the ceftriaxone infusion
Arm/Group | Treatment Sequence AB | Treatment Sequence AC
Number analyzed (Participants) | 5 | 5
ng/mL
  Period 1 | 137,800.0 (10,709.8) | 178,600.0 (34,623.7)
  Period 2 | 143,800.0 (13,103.4) | 169,200.0 (32,782.6)

2. Primary Outcome: Ceftriaxone PK Time to Reach Cmax (Tmax) With (Period 2) and Without (Period 1) SYN-004.
Description: Samples were collected at 0.25 h, 0.5 through 2 h, and 3 through 7 h after the infusion start. Standard deviations may be 0 if all collected T max values occur at the same time.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Sequence AB | Treatment Sequence AC
Number analyzed (Participants) | 5 | 5
hours
  Period 1 | 0.5 (0.0) | 0.5 (0.0)
  Period 2 | 0.5 (0.0) | 0.5 (0.0)

3. Primary Outcome: Ceftriaxone PK Area Under the Concentration-time Curve From Time 0 to the Last Quantifiable Concentration (AUCt) With (Period 2) and Without (Period 1) SYN-004.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Treatment Sequence AB | Treatment Sequence AC
Number analyzed (Participants) | 5 | 5
h*ng/mL
  Period 1 | 464,400.0 (26,884.9) | 656,200.0 (105,257.8)
  Period 2 | 478,800.0 (37,117.4) | 643,800.0 (108,349.9)

ADVERSE EVENTS:
Arm/Group | Low Dose | High Dose
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 4/6 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose (N=6) | High Dose (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Catheter site bruise (General disorders) | 1 | 0
Discomfort (General disorders) | 1 | 0
Feeling cold (General disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators do not see trial results ahead of public disclosure unless it is under CDA. Investigators will not be allowed to publish or disclose any study results prior to sponsor communicating it to the public.